CLINICAL TRIAL: NCT04032951
Title: Evaluation of a Newly Designed 22 Gauge Needle for EUS Guided Tissue Acquisition of Samples for Histologic Examination in Patients With Solid Lesions: A Prospective Two Centers Study
Brief Title: 22 Gauge Needle for EUS Guided Tissue Acquisition of Samples for Histologic Examination
Acronym: EUSFNTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Responsible Party: Principal Investigator, Guido Costamagna, professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10012/14
Record Dates: First submitted 2015-01-19; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Abdominal Neoplasms
Keywords: EUS-guided biopsy
MeSH Terms: conditions — Abdominal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adominal neoplasms patients (Experimental): Patients in whom EUS-FNTA is performed with a novel type of biopsy neede.
  Interventions: Other: Fine Needle Tissue Acquisition

INTERVENTIONS:
Other: Fine Needle Tissue Acquisition — diagnostic
  Other Names: FNTA

SUMMARY:
To determine the yield of tissue biopsy specimen and the diagnostic accuracy of tissue acquisition using a newly developed 22 gauge needle in patients with solid lesions throughout the GI tract.

DETAILED DESCRIPTION:
The use of 22 gauge needle to gather tissue samples under EUS guidance has not been associated with an increased risk, and no major complications have been described so far both for the 22 gauge Procore needle and for standard 22 gauge.20, 21 Potential benefits of this new needle are the possibility of increasing the chance of retrieving tissue specimens for histological examination, with the possibility of increasing the diagnostic accuracy of the procedure saving the need and the cost deriving from on-site cytopathology examination. This may reduce the need to repeat EUS procedures or other more invasive sampling procedures, including surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 and less than 80.
* Presence of a solid lesion within or adjacent of the gastrointestinal tract. In the presence of a cystic component, the solid part of the lesion should be more 75% of the total.
* Absence of an uncorrectable coagulopathy as defined by abnormal prothrombin time (PT) or partial thromboplastin time (PTT) that does not normalize after administration of fresh frozen plasma.
* Informed consent is obtained

Exclusion Criteria:

* Previous biopsy of the lesion with diagnosis of malignancy
* Presence of an uncorrectable coagulopathy as defined by abnormal prothrombin time (PT) or partial thromboplastin time (PTT) that does not normalize after administration of fresh frozen plasma.
* They are unable to understand and/or read the consent form.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
- Yield, as defined by the percentage of patients in whom a histologically interpretable specimen will be retrieved by EUS-FNTA. | intraoperative
  diagnostic accuracy

SECONDARY OUTCOMES:
rate of complications | perioperative
  - The rate of complications, divided in procedural complication (perforation, bleeding) occurring during the procedure and late complications (delayed bleeding, infection) occurring during the post-procedural observational period.

CONTACTS AND LOCATIONS:
Overall Officials: GUIDO COSTAMAGNA, PROF, Study Director — Catholic University of the Sacred Heart
Locations (2):
- Italy (2):
  - ISMETT, Palermo
  - Universita cattolica del sacro cuore, Rome